CLINICAL TRIAL: NCT00936780
Title: Safety and Efficacy of the Infinnium-Core™ Paclitaxel-Eluting Coronary Stent System for the Treatment of Patients With De Novo Coronary Lesions
Brief Title: Infinnium-Core™ Registry for the Treatment of Patients With De Novo Coronary Lesions
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: market demand from paclitaxel to sirolimus drug-eluting stent
Sponsor: Sahajanand Medical Technologies Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC001: V1.1
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Restenosis; Stent thrombosis; Coronary stents; Angioplasty; Drug Eluting Stents (DES)
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Infinnium-Core™ Paclitaxel eluting Coronary Stent (Experimental)
  Interventions: Device: Infinnium-Core™ Paclitaxel eluting Coronary Stent

INTERVENTIONS:
Device: Infinnium-Core™ Paclitaxel eluting Coronary Stent — Infinnium-Core™ Coronary Stent System consisting of the Coronnium® coronary stent (CE approved) having Biodegradable Polymeric Matrix on a Co-Cr alloy Platform. Drug concentration is 1.36 µg/mm2.
  Other Names: Drug Eluting Stent (DES)

SUMMARY:
The primary objective of Infinnium-Core™ Registry is to assess the safety and efficacy of the Infinnium-Core™ Paclitaxel Eluting Coronary Stent System in de novo Coronary Lesions.

DETAILED DESCRIPTION:
Infinnium-Core™ Registry is a multi-centric, prospective study. Approximately 150 patients will be enrolled in the study. Patients will be followed for two years post-procedure.

Data analysis will include all statistically pre assigned 20% patients and all patients who have repeat angiography due to complication. The diabetic patients will be specified as a high risk subset in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Eligible for percutaneous coronary intervention (PCI).
3. Acceptable candidate for CABG.
4. Clinical evidence of ischemic heart disease and/or a positive territorial functional study. Documented stable angina pectoris ((Canadian Cardiovascular Society (CCS) Classification 1,2,3 or 4) or unstable angina pectoris with documented ischemia (Braunwald Class IB-C, IIB-C or IIIB-C), or documented silent ischemia.
5. The target lesion is a single de novo coronary artery lesion with ≥ 50% and < 100% stenosis in one of the major epicardial territories (LAD, LCX or RCA). A second target lesion in another major epicardial vessel could be treated and this second lesion should fit with the inclusion/exclusion criteria and will receive the same type of stent.
6. The target lesion must be covered by one study stent, preferably with a margin of 3 mm on each side of the lesion.
7. The target lesion must be ≤ 37 mm in length by visual estimate.
8. The target reference vessel diameter must be ≥ 2.5 mm and ≤ 3.5 mm.
9. Patient or patient's legal representative has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as notified / approved by the Institutional Review Board/Ethics Committee of the clinical site.

Exclusion Criteria:

1. Female of childbearing potential.
2. Documented left ventricular ejection fraction (LVEF) ≤ 25%.
3. Evidence of an acute Q-wave or non-Q-wave myocardial infarction within 72 hours preceding the index procedure.
4. Known allergies to the following: aspirin, clopidogrel bisulfate (Plavix®, Ceruvin) or ticlopidine (Ticlid®), heparin, paclitaxel, cobalt, chromium, contrast agent (that cannot be adequately pre-medicated).
5. A platelet count <100,000 cells/mm3 or > 700,000 cells/mm3 or a WBC < 3,000 cells/mm3.
6. Acute or chronic renal dysfunction (creatinine > 2.0 mg/dl or > 150 µmol/L).
7. Target vessel has evidence of thrombus.
8. Target vessel is excessively tortuous which makes it unsuitable for proper stent delivery and deployment.
9. Previous bare metal stenting (less than 1 year) anywhere within the target vessel.
10. Previous drug-eluting stenting anywhere within any epicardial vessel
11. The target lesion requires treatment with a device other than PTCA prior to stent placement (e.g., but not limited to, directional coronary atherectomy, excimer laser, rotational atherectomy, etc.)
12. Significant (> 50%) stenosis proximal or distal to the target lesion that might require revascularization or impede run-off.
13. Heavily calcified lesion and/or calcified lesion which cannot be successfully predilated.
14. Target lesion is located in or supplied by an arterial or venous bypass graft.
15. Ostial target lesion.
16. Patient is currently participating in an investigational drug or device study, including its follow-up period.
17. Within 30 days prior to procedure, patient has undergone a previous coronary interventional procedure of any kind.
18. Within 60 days post-procedure, patient requires planned interventional treatment of any non-target vessel. Planned intervention of the target vessel after the index procedure is not allowed.
19. CVA within previous 6 months.
20. Unprotected Left Main (LM) coronary artery disease (stenosis > 50%).
21. In the investigator's opinion, patient has a co-morbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study.
22. Planned surgery within 6 months after the index procedure.
23. Life expectancy less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2008-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | 30 days and 9 month

SECONDARY OUTCOMES:
ANGIOGRAPHIC | 12 months
  In Angiographic outcome measures the Minimal lumen diameter (MLD), % diameter stenosis, In-Stent and In-segment late loss, Proximal late loss, Distal late loss and Binary restenosis rate

CONTACTS AND LOCATIONS:
Locations (7):
- India (7):
  - Bankers Heart Institute, Vadodara, Gujarat
  - Baroda Heart Institute & Research Center, Vadodara, Gujarat
  - CHL Apollo Hospitals,, Indore, Madhya Pradesh
  - CHL Apollo Hospitals, Indore, Madhya Pradesh
  - Government Medical College & Super Speciality Hospital, Nagpur, Maharashtra
  - Arneja Heart Institute, Nagpur, Maharashtra
  - Sri Ramakrishna Heart Foundation & Research Centre, Coimbatore, Tamil Nadu